CLINICAL TRIAL: NCT02362321
Title: Role of Dexamethasone in the Conservative Treatment of Chronic Subdural Hematoma: a Double-blind Randomized Controlled Pilot Study
Brief Title: Role of Dexamethasone in the Conservative Treatment of Chronic Subdural Hematoma
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to serious adverse events
Sponsor: CHU de Quebec-Universite Laval (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PEJ-370
Record Dates: First submitted 2015-02-09; First posted 2015-02-12 (Estimated); Results first posted 2015-02-27 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2016-02

CONDITIONS: Hematoma, Subdural, Chronic
Keywords: [C10.228.140.300.535.450.400.120]
MeSH Terms: conditions — Hematoma, Subdural, Chronic | interventions — Dexamethasone; Adrenal Cortex Hormones; Calcium Dobesilate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexamethasone (Experimental): Participants allocated to the treatment group received a daily dosage of 12mg (4mg three times a day) of dexamethasone for three weeks. Corticosteroid treatment was then tapered off over the next week (8mg for 48 hrs, 4mg for 48 hrs, 2mg for 48 hrs and 1mg for 24 hrs).
  Interventions: Drug: Dexamethasone
- Control (Placebo Comparator): Identical oral capsules filled with lactose were administered to the control (placebo) group for 28 days.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Dexamethasone — Patients received a daily dosage of 12mg (4mg three times a day) of dexamethasone for three weeks. Corticosteroid treatment was then tapered off over the next week (8mg for 48 hrs, 4mg for 48 hrs, 2mg for 48 hrs and 1mg for 24 hrs).
  Other Names: Corticosteroid; Decadron
  Arms: Dexamethasone
Other: Placebo — Identical oral capsules filled with lactose were administered to the control (placebo) group for 28 days.
  Arms: Control

SUMMARY:
Current opinion regarding the use of steroids in the treatment of chronic subdural hematomas are mostly based on observational studies. Here we present data from a prospective randomized pilot study of twenty chronic subdural hematoma (CSDH) patients treated with dexamethasone or placebo for 30 days.

Twenty patients with computed tomography (CT)- or magnetic resonance imaging (MRI)-confirmed CSDH were recruited from a single center and randomized in order to receive dexamethasone or placebo as a conservative treatment. Patients affected to the treatment group received oral dexamethasone 12mg/day for three weeks followed by tapering. These patients were followed for 6 months and the rate of success of conservative treatment versus placebo was measured. Parameters such as hematoma thickness and global impression of change were also compared before and after treatment with chi-square tests. Adverse events and complications were documented.

DETAILED DESCRIPTION:
Patients Recruitment for this single-center double-blind randomized placebo-controlled study was performed between January 2007 and May 2009. Patients were enrolled based on the following inclusion criteria: 18 years and older with evidence of subacute or chronic supratentorial subdural hematoma by CT (computerized tomography) scan or MRI (magnetic resonance imaging) and classified between 0 and 2 using the Markwalder grading scale (17) (Grade 0 for normal neurological status, grade 1 for no neurological deficits but mild symptoms, grade 2 for focal or variable neurological deficits, grade 3 for several focal neurological signs, and grade 4 for comatose). Exclusion criteria included contraindications or intolerance to corticosteroid therapy or patients already undergoing steroid treatment for any other indication, previous neurological surgery up to one year prior to being considered for the study, concomitant cerebral pathology of neoplastic or presumed infectious origin, anticoagulant therapy that could not be stopped for 6 months and refusal to participate in the study. If at any time, patients developed a sudden increase in hematoma volume, a midline displacement of greater than 1cm or a deterioration of their level of consciousness, they were removed from the conservative study protocol in order to undergo surgery.

This study was approved by the research ethics board at Centre Hospitalier Universitaire (CHU) de Quebec. Written and fully informed consent was obtained from each participant.

Randomization Allocation to each group was done in a 1:1 ratio with block sizes ranging from 4 to 6, to one of the two arms ; a treatment arm in which participants received dexamethasone according to the protocol, and a control group in which they received placebo. Randomization was performed via a web-based service by a pharmacist, which was not involved in any other part of the study. Both investigators and participants were blind to treatment allocation.

Treatment Participants allocated to the treatment group received a daily dosage of 12mg (4mg three times a day) of dexamethasone for three weeks. Corticosteroid treatment was then tapered off over the next week (8mg for 48 hrs, 4mg for 48 hrs, 2mg for 48 hrs and 1mg for 24 hrs). Identical oral capsules filled with lactose were administered to the control (placebo) group for 28 days. Participants were returned at home with blister packs containing their medication for each day of the trial and were asked to return empty packs to ensure compliance with the assigned treatment. The treatment (placebo or dexamethasone) was discontinued if a patient required surgical drainage of its hematoma or suffered from significant side effects.

Evaluation and follow-up The primary outcome of this pilot study was to determine the efficacy of dexamethasone as compared with placebo in reducing the rate of surgical intervention for CSDH graded 0 to 2 on the Markwalder grading scale (Grade 0 for normal neurological status, grade 1 for no neurological deficits but mild symptoms, grade 2 for focal or variable neurological deficits, grade 3 for several focal neurological signs, and grade 4 for comatose).

Eligible patients who consented for the study underwent the routine standard of care. This included 1) a complete medical history review and neurological physical exam ; 2) head computerized tomography (CT) or MRI with measurement of maximal hematoma thickness (in mm), midline shift ; 3) and a check of blood and vital parameters. In addition, patients were asked to complete detailed questionnaires measuring symptoms typically associated with subdural hematomas.

Follow-up appointments were scheduled 2 weeks, 1, 2 and 6 months after initiation of treatment. At each visit, the three components of the clinical evaluation described above were repeated. Moreover, a seven point categorical scale was used to evaluate patient's global impression of change relative to the initial state (unchanged , very much improved, much improved, minimally improved, minimally worse, much worse, very much worse). Treatment-related side effects were also inquired about and collected.

The rate of success of conservative management was defined as the percentage of patients not requiring surgery in each treatment group during the 6 months following enrollment. Radiological progression of the hematoma in terms of thickness and magnitude of midline shift, hematoma-related symptoms and medication-related side effects were carefully collected.

Statistical analyses Demographical characteristics, baseline neurological status and hematoma size and location were compared for both groups using a Mann-Whitney test for continuous variable and a χ2 test for categorical variables.

To compare the rate of success, a categorical frequency comparison with the Fisher's exact test was used. For the other outcome measures we used Mann-Whitney U test and Student's t-test for normally distributed variables and χ2 or Fisher's exact test for categorical frequencies. All statistical tests were done with the Statistical package for Social Sciences software version 16.0 and the significance threshold was set at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* evidence of subacute or chronic supratentorial subdural hematoma by CT (computerized tomography) scan or MRI (magnetic resonance imaging)
* classified between 0 and 2 using the Markwalder grading scale

Exclusion Criteria:

* contraindications or intolerance to corticosteroid therapy
* patients already undergoing steroid treatment for any other indication
* previous neurological surgery up to one year prior to being considered for the study
* concomitant cerebral pathology of neoplastic or presumed infectious origin
* anticoagulant therapy that could not be stopped for 6 months
* refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-01; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dexamethasone | Control
Started | 10 | 10
Completed | 6 | 10
Not Completed | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexamethasone | Control | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 3 | 4
  >=65 years | 9 | 7 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.3 (6.3) | 69.4 (8.8) | 70.9 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 10 | 8 | 18
Region of Enrollment [Number; unit: participants]
  Canada | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Rate of Need for Surgery Drainage
Description: The rate of success of conservative management was defined as the number of patients not requiring surgery in each treatment group during the 6 months following enrollment.
Time Frame: Within 6 months
Measure: Number; unit: participants
Arm/Group | Dexamethasone | Control
Number analyzed (Participants) | 10 | 10
participants | 9 | 7

ADVERSE EVENTS:
Arm/Group | Dexamethasone | Control
Serious Adverse Events (participants affected / at risk) | 8/10 | 2/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dexamethasone (N=10) | Control (N=10)
Hyperglycemia (Endocrine disorders) | 4 (4) | 1 (1)
High pressure (Cardiac disorders) | 1 (1) | 0 (0)
Pulmonary embolus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cellulitis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Suicide (Psychiatric disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No